CLINICAL TRIAL: NCT06015139
Title: Comparison of the Effectiveness of Positioning Device Cotton Roll-coated Viscoelastic Polymer Pads Versus Viscoelastic Polymer Pads for Preventing Pressure Injuries in Patients Undergoing Lumbar Spine Surgery
Brief Title: Preventing Pressure Injuries in Patients Undergoing Lumbar Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Taiwan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yu, Hsing-Sheng, Principal Investigator, Central Taiwan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 游行盛
Record Dates: First submitted 2023-07-03; First posted 2023-08-29 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Pressure Injury
Keywords: pressure injury; positioning devices; prophylactic
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- viscoelastic polymer pads (Active Comparator): while the control group used a Relton-Hall prone frame with a viscoelastic polymer pads
  Interventions: Device: viscoelastic polymer pads
- cotton roll-coated viscoelastic polymer pads (Experimental): The experimental group used a Relton-Hall prone frame with cotton roll-coated 3 cm viscoelastic polymer pads
  Interventions: Device: cotton roll-coated viscoelastic polymer pads

INTERVENTIONS:
Device: cotton roll-coated viscoelastic polymer pads — relton-hall frame cotton roll-coated viscoelastic polymer pads
  Arms: cotton roll-coated viscoelastic polymer pads
Device: viscoelastic polymer pads — relton-hall frame viscoelastic polymer pads
  Arms: viscoelastic polymer pads

SUMMARY:
Background：Pressure injuries (PI) are one of the common comorbidities in surgery, meaning PI that occurs immediately after surgery or within hours to 3 days after surgery. The incidence of PI in spine surgery is about 5% ~ 66%.

Purpose：Comparison of the difference in pressure injury rates positioning device cotton roll-coated viscoelastic polymer pads versus viscoelastic polymer pads for pressure injuries undergoing lumbar spine surgery Methods：This experimental study used a split-body design with random assignment to compare the pressure-reducing effects of different materials on a patient's body contact points with a positioning device. The experimental group used a Relton-Hall prone frame with cotton roll-coated 3 cm viscoelastic polymer pads, while the control group used a Relton-Hall prone frame with a viscoelastic polymer pads.

DETAILED DESCRIPTION:
The study focuses on patients undergoing lumbar surgery in a hospital in a certain area of northern Taiwan, with an intended recruitment of 50 participants randomized into experimental and control groups. The study will use the Pressure Injury grading system developed by the National Pressure Injury Advisory Panel to assess the severity of pressure injuries at pre-operation, immediate post-operation, 30 minutes post-operation, 24 hours post-operation, and 48 hours post-operation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving lumbar nerve decompression combined with internal fixation and bone fusion.
2. Use the positioning device Relton-Hall rack in prone position.
3. The operation time is more than 2.5 hours.
4. The surgical anesthesia is general anesthesia.
5. Routine surgery registered on the surgery schedule.
6. Before the operation, the skin was intact and there was no pressure injury.

Exclusion Criteria:

1. Emergency lumbar surgery patients.
2. Under the age of 18.
3. The operation time is less than 2.5 hours.
4. Preoperative skin incompleteness (obviously there is chest and iliac crest crush phenomenon).
5. Percutaneous minimally invasive disc herniation decompression (percutaneous endoscopic lumbar disc, PELD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Comparing two kinds of decompression materials, the incidence of Pressure Injury in lumbar patients after surgery | immediate post-operation, 30 minutes post-operation, 24 hours post-operation, and 48 hours post-operation
  The four parts of the patient's body in contact with the positioning device (left chest, left iliac crest and right chest, right iliac crest) were randomly divided into an experimental group or a control group, and the decompression effect of different materials on positioning the device on the patient's body was compared; the experiment The group used the positioning device Relton-Hall prone frame cotton roll to cover the 3 cm fat pad, and the control group used the Relton-Hall prone frame fat pad.
  The severity of PI in the experimental and control groups was assessed and measured according to the pressure injury grading developed by the National Pressure Injury Advisory Committee. After surgery, return the patient from the prone position to the supine position. Immediately after the operation, 24 hours and 48 hours after the operation, observe the occurrence of pressure injury in the experimental group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Ying Dai, Study Director — advising professor
Locations (1):
- Dachien Hospital, Miaoli, Gongjing Rd, Taiwan

DOCUMENTS (2):
  • Study Protocol: Proposal (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT06015139/Prot_000.pdf
  • Study Protocol and Informed Consent Form: Subject Consent (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT06015139/Prot_ICF_001.pdf